CLINICAL TRIAL: NCT03378648
Title: A First In Human Randomised, Double-Blind, Placebo-Controlled Study Of Single Ascending Doses In Healthy Male Volunteers And Repeated Ascending Dose In Asthmatic Patients Followed By A 3-Way Cross-Over, Placebo-Controlled, Single-Dose In Copd Patients To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of CHF6366
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Dose in Healthy Volunteers, Repeat Doses in Asthmatic Patients and of Single Dose in COPD Patients of CHF6366
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06366AA1-01; 2015-005551-27 (EudraCT Number)
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Part 1 alternating cross-over design
  Part 2 parallel group design
  Part 3 3-way cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 double-blind
  Part 2 double-blind
  Part 3 placebo-controlled (double-blind), active-controlled (open labelled)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHF6366 active (Experimental)
  Interventions: Drug: CHF6366
- CHF6366 (Placebo Comparator)
  Interventions: Drug: Placebo CHF6366
- Comparator (Active Comparator)
  Interventions: Drug: umeclidinium bromide and vilanterol trifenatate

INTERVENTIONS:
Drug: CHF6366 — Drug: CHF6366 (Part 1 - SAD) Single doses of CHF6366 at each period (for up to 3 periods per subject)
  Drug: CHF6366 (Part 2 - MAD) Once daily doses of CHF6366 for 7 days
  Drug: CHF6366 (Part 3) Single dose of CHF6366
  Arms: CHF6366 active
Drug: Placebo CHF6366 — Drug: Placebo (Part 1 - SAD) Single doses of placebo matching CHF6366 at each period (for up to 3 periods per subjects)
  Drug: Placebo (Part 2 - MAD) Once daily dose of placebo matching CHF6366 for 7 days
  Drug: Placebo (Part 3) Single dose of placebo matching CHF6366
  Arms: CHF6366
Drug: umeclidinium bromide and vilanterol trifenatate — Part 3 Single dose
  Arms: Comparator

SUMMARY:
CHF6366 is a novel bifunctional compound displaying both muscarinic receptor antagonist and β2-adrenergic receptor agonist properties (MABA), with the potential to deliver optimal bronchodilation after inhalation dosing via two validated mechanisms in one molecule.

The study will consist of three parts:

Part 1 will consit of two cohorts of healthy male subjects to assess the safety, tolerability and pharmacokinetics of Single Ascending Dose (SAD) of CHF 6366

Part 2 will consist of four cohorts of asthmatic subjects to assess the saftey, tolerability and pharmacokinetics of Multiple Ascending Dose (MAD) of CHF6366

Part 3 will consist of one cohort of COPD patients to asess safety, tolerability of a single dose of CHF6366 in an active and placebo controlled design

ELIGIBILITY:
Inclusion Criteria:

Part 1

* male subjects aged 18-55 years inclusive;
* healthy subjects based on medical evaluation including medical history,physical examination, laboratory tests and cardiac testing
* Body Mass Index (BMI) between 18.5 and 32.0 kg/m2 extremes inclusive
* Non- or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking > 1 year;
* Good physical and mental status, determined on the basis of the medical history and a general clinical examination;
* Lung function equal to or more than 80% of predicted normal value and FEV1/FVC ratio > 0.70;

Part 2

* Adult male and female subjects aged 18 to 75 years
* Clinical diagnosis of mild persistent asthma
* FEV1 reversibility of ≥ 12% or 200 ml over the baseline value starting within 30 mins after inhalation of 400 micrograms of salbutamol
* Patients who are otherwise healthy as determined by medical history, physical examination, 12-lead ECG findings

Part 3

* Male aged between 40 and 75 years
* Stable patients with a post-bronchodilator 40% ≤ FEV1 < 80% of the predicted normal value, post-bronchodilator FEV1/FVC < 0.7 with salbutamol
* Current smokers and ex-smokers
* Response to ipratropium bromide defined as an increase in FEV1 of > 7 % starting 30 minutes after inhalation of 80 micrograms ipratropium bromide
* Response to salbutamol defined an increase in FEV1 of > 7 % starting 15 minutes to 30 min following inhalation of 400 micrograms salbutamol MDI

Exclusion Criteria:

Part1

* Any clinically relevant abnormabilites and/or uncontrolled diseases
* Abnormal laboratory values
* Recent respiratory tract infection
* Hypersensitivity to the drug excipients
* Positive serology results
* Positive cotinine, alcohol, drug of abuse tests

Part 2

* Pregnant and/or breast-feeding women
* Subjects with a medical history or current diagnosis of COPD or any other pulmonary disease other than asthma
* Subjects who have cardiovascular condition
* Clinically significant laboratory abnormalities
* Subject with serum potassium level below the lower limit of the laboratory reference range
* History of alcohol, substance or drug abuse
* Hypersensitivity to the drug excipients

Part 3

* Female patients
* Current diagnosis of asthma or allergic rhinitis or other atopic disease
* Recent COPD exacerbations or a lower respiratory tract infection
* Hypersensitivity to drug excipients;
* Abuse of substance or drug t or with a positive urine drug screen
* Unstable concurrent disease
* Subjects who have cardiovascular condition
* Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease
* Patients with serum potassium levels below the lower limit of the laboratory normal range

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Part 1 from Day 1 until day 3, Part 2 from Day 1 until day 8, Part 3 from Day 1 until Day 3 (per each period)
Vital signs | Part 1 from Day 1 until Day 3, Part 2 from Day 1 until day 8, Part 3 from Day 1 until Day 3 (per each period)
  Systolic, diastolic Blood Pressure
Change in Holter ECG parameters | Part 1 from Day 1 until Day 3, Part 2 from Day 1 until day 8, Part 3 from Day 1 until Day 3 (per each period)
  HR, PR, QRS, QTcF, QT
Change in Holter parameters | Part 1 from Day 1 until Day 3, Part 2 from Day 1, until Day 8, Part 3 from Day 1 until Day 3(per each period)
Change in FEV1 | Part 1 drom Day 1 until Day 3, Part 2 from Day 1 until Day 8
  Forced expiratory capacity in the first second
Change in Laboratiry parameters | Part 1 Day -1 and Day 3, Part 2 Day -2 and Day 8, Part 3 Day -1 and Day 2
  clinical chemistry, haematology and urinanalysis
Change in serum potassium level | Part 1 Day 1, Part 2 Day 1 and Day 7, Part 3 Day 1

SECONDARY OUTCOMES:
Area under the plasma concentration vs time curve | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
Peak plasma concentration (Cmax) | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
  maximum plasma concentration of CHF6366
Time to reach the maximum plasma concentration (tmax) | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
Elimination half-life (t1/2) | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
Clearance (CL/F) | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
Volume of distribution (Vz/F) | Part 1 Day 1 until Day 3, Part 2 Day 1 , Part 3 Day 1 until Day 3 (per each period)
Area under the plasma concentration vs time curve during selected dosing interval | Part 2 Day 7
Peak plasma concentration during selected dosing (Cmaxss) | Part 2 Day 7
Value of minimum plasma concentration post dosing at selected dosing interval (Cminss) | Part 2 Day 7
Time of minimum plasma concentration post dosing at selected dosing interval (Tminss) | Part 2 Day 7
Time to reach the maximum plasma concentration at selected dosing interval(tmaxss) | Part 2 Day 7
Clearance at selected dosing interval (CL/Fss) | Part 2 Day 7
Volume of distribution at selected dosing interval (Vz/Fss) | Part 2 Day 7
Accumulation ratio (Rac) | Part 2 Day 7
Steady state concentration (Css) | Part 2 Day 7
Urinary excretion (Ae) | Part 1 from Day 1 until Day 3, Part 2 Day 1 and Day 7, Part 3 from Day 1 until Day 3 (per each period)
fraction excreted (fe) | Part 1 from Day 1 until Day 3, Part 2 Day 1 and Day 7, Part 3 from Day 1 until Day 3 (per each period)
Clearance (CLr) | Part 1 from Day 1 until Day 3, Part 2 Day 1 and Day 7, Part 3 from Day 1 until Day 3 (per each period)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CCD-06366AA1-01